CLINICAL TRIAL: NCT05682768
Title: Buttressed Pancreatico-Gastrostomy for Soft Pancreas With Small Pancreatic Duct Diameter in Whipple Procedure. A Retrospective Cohort Study
Brief Title: Buttressed Pancreatico-Gastrostomy for Soft Pancreas With Small Diameter Pancreatic Duct in Whipple Procedure
Status: Completed | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Abdallah Mohamed Taha Aly, Assistant Professor, South Valley University
Other Study IDs: SVU-MED-SUR011-4-22-10-465
Record Dates: First submitted 2022-12-26; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Pancreatic Fistula
Keywords: Cancer pancreas; Pancreaticoduodenectomy; Pancreaticogastrostomy
MeSH Terms: conditions — Pancreatic Fistula; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with cancer pancreas with soft pancreas and non-dilated pancreatic duct
  Interventions: Procedure: Duct to Mucosa Pancreatico-Gastrostomy with trans-pancreatic transverse mattress U- Shaped sutures

INTERVENTIONS:
Procedure: Duct to Mucosa Pancreatico-Gastrostomy with trans-pancreatic transverse mattress U- Shaped sutures — Adding suporting sutures between th posterior gastric wall and ancreatic stump in whipple procedure, the sutures are Duct to Mucosa Pancreatico-Gastrostomy with trans-pancreatic transverse mattress U- Shaped sutures.
  Other Names: Buttressing sutures

SUMMARY:
Post-operative pancreatic fistula after Pancreaticoduodenectomy procedure, is still a major complication that might be affected by pancreatic stump reconstruction technique. More than 60 techniques were published in literature. Soft pancreas and small pancreatic duct size were major risk factors for post-operative pancreatic fistula. Supporting Duct to Mucosa Pancreatico-Gastrostomy with trans-pancreatic transverse mattress U- Shaped sutures is a new and safe technique for decreasing the risk of post-operative pancreatic fistula in high-risk patients.

DETAILED DESCRIPTION:
Post-operative pancreatic fistula after Pancreaticoduodenectomy procedure, is still a major complication that might be affected by pancreatic stump reconstruction technique. More than 60 techniques were published in literature. Soft pancreas and small pancreatic duct size were major risk factors for post-operative pancreatic fistula. Supporting Duct to Mucosa Pancreatico-Gastrostomy with trans-pancreatic transverse mattress U- Shaped sutures is a new and safe technique for decreasing the risk of post-operative pancreatic fistula in high-risk patients.

The authors used this technique in pancreato-gastrostomy. Data were collected, tabulated and analyzed to evaluate the new technique and its impact on the incidence of post-operative pancreatic fistula.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with resectable cancer head pancreas.
* Soft Pancreas.
* Small pancreatic duct diameter.

Exclusion Criteria:

* Unresectable cancer pancreas.
* Non soft pancreas.
* Dilated pancreatic duct.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with soft pancreas and pancreatic duct diameter ≤ 5 mm (15 Fr), who underwent the classic pancreaticoduodenectomy (Whipple) procedure for cancer pancreas. Supporting pancreatico-gastrostomy with buttressing sutures was used. It is an anastomotic modification by supporting it with trans-pancreatic and full-thickness gastric wall transverse mattress U- Shaped sutures to fix the posterior gastric wall envelope around the pancreatic stump, to alleviate any tension on the Pancreatico-Gastrostomy sutures.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
Post operative Pancreatic Fistula | up to 5 days (from time of surgery to time of detection of post-operative pancreatic fistula)
  Detection of chemical or clinical pancreatic fluid discharge after post-operative day 3.

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah M Taha, MD, Principal Investigator — South Valley University, Faculty of Medicine
Locations (1):
- Qena Faculty of Medicine, South Valley University Hospitals, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No
Study Protocol Statistical Analysis Plan

REFERENCES:
- [Background] Callery MP, Pratt WB, Vollmer CM Jr. Prevention and management of pancreatic fistula. J Gastrointest Surg. 2009 Jan;13(1):163-73. doi: 10.1007/s11605-008-0534-7. Epub 2008 May 22. PMID 18496727
- [Background] Lai EC, Lau SH, Lau WY. Measures to prevent pancreatic fistula after pancreatoduodenectomy: a comprehensive review. Arch Surg. 2009 Nov;144(11):1074-80. doi: 10.1001/archsurg.2009.193. PMID 19917946
- [Background] Osada S, Imai H, Sasaki Y, Tanaka Y, Nonaka K, Yoshida K. Reconstruction method after pancreaticoduodenectomy. Idea to prevent serious complications. JOP. 2012 Jan 10;13(1):1-6. PMID 22233940
- [Background] Callery MP, Pratt WB, Kent TS, Chaikof EL, Vollmer CM Jr. A prospectively validated clinical risk score accurately predicts pancreatic fistula after pancreatoduodenectomy. J Am Coll Surg. 2013 Jan;216(1):1-14. doi: 10.1016/j.jamcollsurg.2012.09.002. Epub 2012 Nov 2. PMID 23122535
- [Background] Schmidt CM, Choi J, Powell ES, Yiannoutsos CT, Zyromski NJ, Nakeeb A, Pitt HA, Wiebke EA, Madura JA, Lillemoe KD. Pancreatic fistula following pancreaticoduodenectomy: clinical predictors and patient outcomes. HPB Surg. 2009;2009:404520. doi: 10.1155/2009/404520. Epub 2009 May 18. PMID 19461951
- [Background] Lermite E, Pessaux P, Brehant O, Teyssedou C, Pelletier I, Etienne S, Arnaud JP. Risk factors of pancreatic fistula and delayed gastric emptying after pancreaticoduodenectomy with pancreaticogastrostomy. J Am Coll Surg. 2007 Apr;204(4):588-96. doi: 10.1016/j.jamcollsurg.2007.01.018. Epub 2007 Mar 2. PMID 17382217
- [Background] Bassi C, Falconi M, Molinari E, Salvia R, Butturini G, Sartori N, Mantovani W, Pederzoli P. Reconstruction by pancreaticojejunostomy versus pancreaticogastrostomy following pancreatectomy: results of a comparative study. Ann Surg. 2005 Dec;242(6):767-71, discussion 771-3. doi: 10.1097/01.sla.0000189124.47589.6d. PMID 16327486